CLINICAL TRIAL: NCT02918071
Title: A Multicenter, Open-Label, Functionality, Reliability and Performance Study of a Single-Use Auto-Injector With Home-administered Subcutaneous Benralizumab in Adult Patients With Severe Asthma (GRECO)
Brief Title: Study to Assess Functionality, Reliability, and Performance of a Single-Use Auto-Injector With Benralizumab Administered at Home
Acronym: GRECO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00031
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Asthma,; Bronchial Diseases,; Respiratory Tract Diseases,; Lung Diseases,; Obstructive Lung Diseases,; Benralizumab
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm Benralizumab (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks

SUMMARY:
The purpose of the study is to assess functionality, performance, and reliability of an single-use auto-injector (AI) with benralizumab administered subcutaneously (SC) in an at-home setting reported by the patient or caregiver, and to confirm the safety and clinical benefit of benralizumab administration in asthma patients with severe asthma

ELIGIBILITY:
Inclusion criteria

* Written informed consent for study participation must be obtained prior to any study related procedures being performed and according to international guidelines and/or applicable European Union (EU) guidelines
* Male and female patients aged 18 to 75 years of age at the time of Visit 1
* Patient or caregiver must be willing and able to self-administer the Investigational product (IP). Caregiver must be age of consent or older at the time of Visit 1, if applicable
* Weight of ≥40 kg
* Evidence of asthma as documented by airway reversibility (FEV1 ≥12% and 200 ml) demonstrated at Visit 1 or 1A or Visit 2
* Documented history of current treatment with Inhaled corticosteroids (ICS) and Long-acting β2 agonists (LABA). The ICS and LABA can be parts of a combination product or given by separate inhalers. The ICS dose must be greater than or equal to 500 μg/day fluticasone propionate dry powder formulation or equivalent daily. For ICS/LABA combination preparations, both the mid- and high-strength maintenance doses approved in the local country will meet this ICS criterion. Additional asthma controller medications (e.g., Leukotriene receptor antagonists (LTRAs), tiotropium, theophylline, oral corticosteroids) are allowed
* Pre-bronchodilator (pre-BD) FEV1 of >50% predicted normal at Visit 1 or 1A or Visit 2
* Not well controlled asthma as documented by either: An Asthma Control Questionnaire 6 (ACQ6 ) ≥1.5 OR; A peak flow of 60-80% predicted OR; One or more exacerbation that required oral or systemic corticosteroids in the previous year

Exclusion criteria:

* Clinically important pulmonary disease other than asthma (eg, active lung infection, COPD (Chronic obstructive pulmonary disease), bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome)
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could: Affect the safety of the patient throughout the study; Influence the findings of the studies or their interpretations; Impede the patient's ability to complete the entire duration of study
* Known history of allergy or reaction to the IP formulation
* History of anaphylaxis to any biologic therapy
* History of Guillain-Barré syndrome
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening
* Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T. Ferguson, MD, PC, Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (23):
- United States (14):
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Westminster, California
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Canton, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Boerne, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
- Canada (9):
  - Research Site, Sherwood Park, Alberta
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Kanata, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4092&filename=d3250c00031-csp-v-1_REDACTED.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4092&filename=d3250c00031-sap-ed-2_REDACTED.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 participants receive treatment with benralizumab 30 mg at every 4 weeks schedule.
Groups:
- Benra 30 mg: Benralizumab administered subcutaneously every 4 weeks
Period: Overall Study
Arm/Group | Benra 30 mg
Started | 121
Completed | 118
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full analysis set
  Years | 48.5 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    Female | 77
    Male | 44
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full analysis set
  Participants
    White | 97
    Black or African American | 14
    Asian | 9
    Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients/Caregivers Who Successfully Administered Benralizumab 30 mg Subcutaneously (SC) by Injection With an AI Device at Home
Description: Patients who are still in the study is defined as patients who had been treated for the specified timepoint. A successful administration is defined as an injection completed, an answer of "Yes" to all 5 questions in the Questionnaire, and adequately passed the visual inspection and function tests.
Time Frame: Week 12, Week 16, Week 12 and 16
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Benra 30mg: Benralizumab administered subcutaneously every 4 weeks
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
Participants
  Week 12: number analyzed (Participants) | 116
  Week 12 | 113
  Week 16: number analyzed (Participants) | 116
  Week 16 | 112
  Week 12 and 16: number analyzed (Participants) | 116
  Week 12 and 16 | 108
Statistical Analysis 1: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); percentage = 97.4, 95% CI 2-sided [92.63 to 99.46] — Percentage of patients successfully administered benralizumab with an AI at home (Week 12)
Statistical Analysis 2: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 16); Percentage = 96.6, 95% CI 2-sided [91.41 to 99.05] — Percentage of patients who successfully administered benralizumab with an AI at home (Week 16)
Statistical Analysis 3: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12 and 16); Percentage = 93.1, 95% CI 2-sided [86.86 to 96.98] — Percentage of patients who successfully administered benralizumab with an AI at home (Week 12 and 16)

2. Primary Outcome: Number of Returned AI Devices Used to Administer Benralizumab at Home That Have Been Evaluated as Functional
Description: AI evaluated as functional is defined as the device having adequately passed the visual inspection and function tests.
Time Frame: Week 12, Week 16
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Count of Units; unit: Auto-injector
Units Other Than Participants: Auto-injector
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
Number analyzed (Auto-injector) | 234
Auto-injector
  Week 12: number analyzed (Participants) | 116
  Week 12: number analyzed (Auto-injector) | 117
  Week 12 | 114
  Week 16: number analyzed (Participants) | 116
  Week 16: number analyzed (Auto-injector) | 117
  Week 16 | 113
Statistical Analysis 1: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); Percentage = 97.4, 95% CI 2-sided [92.69 to 99.47] — Percentage of patients returned functional AI administered at home (Week 12)
Statistical Analysis 2: Comparison: Benra 30mg; Test type: Other; Clopper Pearson Exact CI; One sample confidence interval (Week 16); Percentage = 96.6, 95% CI 2-sided [91.48 to 99.06] — Percentage of patients returned functional AI administered at home (Week 16)

3. Primary Outcome: Number of AI Devices Used to Administer Benralizumab at Home or in the Clinic and Have Been Reported as Malfunctioning (Product Complaints)
Description: Number (%) of AI used to administer benralizumab at home or in the clinic and have been reported as malfunctioning (Product Complaints). The percentage is calculated based on AI dispensed for patients who were treated for the specific time point. This excludes AIs dispensed but never used for the treatment or the device not returned for evaluation.
Time Frame: Weeks 0, 4, 8, 12, 16, 0 to 8, 12 to 16, and 0 to 16
Population: Number of Units analyzed per row represents number of auto-injector used at each time point.
Measure: Count of Units; unit: Auto-injector
Units Other Than Participants: Auto-injector
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
Number analyzed (Auto-injector) | 595
Auto-injector
  Week 0: number analyzed (Auto-injector) | 121
  Week 0 | 0
  Week 4: number analyzed (Auto-injector) | 121
  Week 4 | 1
  Week 8: number analyzed (Auto-injector) | 119
  Week 8 | 1
  Week 12: number analyzed (Auto-injector) | 117
  Week 12 | 3
  Week 16: number analyzed (Auto-injector) | 117
  Week 16 | 4
  Week 0 to Week 8: number analyzed (Auto-injector) | 361
  Week 0 to Week 8 | 2
  Week 12 to Week 16: number analyzed (Auto-injector) | 234
  Week 12 to Week 16 | 7
  Week 0 to Week 16 | 9
Statistical Analysis 1: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0); Percentage = 0.0, 95% CI 2-sided [0.00 to 3.00] — Percentage of mulfunctioning AI used to administer benralizumab at home or clinic (Week 0)
Statistical Analysis 2: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 4); Percentage = 0.8, 95% CI 2-sided [0.02 to 4.52] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 4)
Statistical Analysis 3: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 8); Percentage = 0.8, 95% CI 2-sided [0.02 to 4.59] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 8)
Statistical Analysis 4: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); Percentage = 2.6, 95% CI 2-sided [0.53 to 7.31] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 12)
Statistical Analysis 5: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 16); Percentage = 3.4, 95% CI 2-sided [0.94 to 8.52] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 16)
Statistical Analysis 6: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0 to 8); Percentage = 0.6, 95% CI 2-sided [0.07 to 1.99] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 0 to 8)
Statistical Analysis 7: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12 to 16); Percentage = 3.0, 95% CI 2-sided [1.21 to 6.07] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 12 to 16)
Statistical Analysis 8: Comparison: Benra 30mg; Test type: Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0 to 16); Percentage = 1.5, 95% CI 2-sided [0.69 to 2.85] — Percentage of malfunctioning AI used to administer benralizumab at home or clinic (Week 0 to 16)

4. Secondary Outcome: Change From Baseline in Mean Asthma Control Questionnaire-6 (ACQ-6) Score
Description: The effect of benralizumab on asthma control metrics in terms of change from baseline in mean Asthma Control Questionnaire-6 (ACQ-6) score. ACQ-6 score is defined as the average of the first 6 items of the ACQ questionnaire on symptoms, activity limitations, and rescue medication. Baseline is defined as the last non-missing observation prior to the first dose of study treatment. ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Smaller score indicates better controlled asthma.
Time Frame: Week 0 (baseline) and weeks 4, 8, 12, 16, 20
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
Scores on a scale
  Week 4 | -0.63 (0.99)
  Week 8: number analyzed (Participants) | 119
  Week 8 | -0.91 (1.05)
  Week 12: number analyzed (Participants) | 117
  Week 12 | -1.07 (1.02)
  Week 16: number analyzed (Participants) | 116
  Week 16 | -1.13 (1.06)
  Week 20: number analyzed (Participants) | 116
  Week 20 | -1.04 (1.08)

5. Secondary Outcome: The Pharmacokinetics (PK) of Benralizumab in the Terms of PK Parameters: Serum Concentration of Benralizumab
Description: Mean PK Concentration at each visit
Time Frame: Baseline, Week 8, Week 20, and Week 28
Population: PK analysis set - include all patients who had at least one quantifiable serum PK observation post first dose of Benralizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
ng/mL
  Baseline | NA (NA) — Value is less than lower limit of quantification
  Week 8: number analyzed (Participants) | 118
  Week 8 | 698.18 (186.455)
  Week 20: number analyzed (Participants) | 115
  Week 20 | 787.51 (280.788)
  Week 28: number analyzed (Participants) | 117
  Week 28 | 62.86 (469.359)

6. Secondary Outcome: The Pharmacodynamics of Benralizumab in the Terms of Peripheral Blood Eosinophil Levels
Description: Blood eosinophil counts by timepoint
Time Frame: Baseline, Week 20, and Week 28
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Median (Inter-Quartile Range); unit: cells/ uL
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
cells/ uL
  Baseline | 230 [150 to 360]
  Week 20: number analyzed (Participants) | 118
  Week 20 | 20 [10 to 30]
  Week 28: number analyzed (Participants) | 115
  Week 28 | 20 [10 to 50]

7. Secondary Outcome: The Immunogenicity of Benralizumab in the Terms of Anti-drug Antibodies (ADA)
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive is defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive
Time Frame: Baseline until Week 28
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Number; unit: Participants
Arm/Group | Benra 30mg
Number analyzed (Participants) | 121
Participants
  Positive at any visit | 9
  Base- and Post-baseline Positive: number analyzed (Participants) | 120
  Base- and Post-baseline Positive | 0
  Only post-baseline positive: number analyzed (Participants) | 120
  Only post-baseline positive | 9
  Only baseline positive | 0
  Persistently Positive: number analyzed (Participants) | 120
  Persistently Positive | 8
  Transiently Positive: number analyzed (Participants) | 120
  Transiently Positive | 1

ADVERSE EVENTS:
Time Frame: 28 weeks.
Description: Adverse events were collected from the time the patient signed the informed consent, throughout the treatment period and including the follow-up period (through Week 28).
  Serious adverse events were recorded from the time of informed consent.
Arm/Group | Benra 30 mg
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 1/121
Other Adverse Events (participants affected / at risk) | 45/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=121)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=121)
Seasonal allergy (Immune system disorders) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 10 (11)
Viral upper respiratory tract infection (Infections and infestations) | 18 (22)
Headache (Nervous system disorders) | 8 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT02918071/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT02918071/SAP_001.pdf